CLINICAL TRIAL: NCT05020431
Title: Detection of Type I Collagen Fragments in the Gingival Crevicular Fluid and Saliva During Orthodontic Tooth Movement
Brief Title: Type I Collagen Fragments in the GCF and Saliva During OTM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Omar Tareq, Principal Investigator, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Collagen Fragments ICTP, CTX.
Record Dates: First submitted 2021-08-22; First posted 2021-08-25 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Collagen Degeneration
Keywords: Orthodontic tooth movement(OTM);; Type I collagen fragments(ICTP, CTX);; Gingival crevicular fluid (GCF);; Saliva.
MeSH Terms: conditions — Xanthomatosis, Cerebrotendinous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm (Experimental): One arm nonrandomized clinical trial
  Interventions: Other: Biological measuring of collagen fragments biomarker during orthodontic tooth movement

INTERVENTIONS:
Other: Biological measuring of collagen fragments biomarker during orthodontic tooth movement — Biological measure the levels of type I collagen fragments ICTP and CTX levels in the GCF and saliva during initial leveling and alignment in adolescent patients treated with fixed orthodontic appliances.

SUMMARY:
Investigate the levels of type I Collagen fragments ICTP and CTX in GCF and saliva during initial leveling and alignment of the teeth in a sample of adolescents undergoing orthodontic treatment.

DETAILED DESCRIPTION:
Type I Collagen fragments ICTP (cross-linked carboxyterminal telopeptide of type 1 collagen) and CTX (C-terminal cross-linked telopeptide of type I collagen) are specific bone resorption biomarkers released in the circulation after osteoclastic bone resorption and collagen degradation and were found to be released in gingival crevicular fluid (GCF) and saliva during metabolic bone diseases and active periodontitis. So the aim of the study is to investigate the levels of ICTP and CTX in GCF and saliva during initial leveling and alignment of the teeth in a sample of adolescents undergoing orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* The age ranges from 13-18 years old.
* Good oral hygiene.
* Clinical gingival health on the intact periodontium.
* Permanent dentition.
* Moderate crowding.
* Non-extraction treatment plan. If extraction of teeth is required, the treatment plan should allow for postponing extraction after sample collection.

Exclusion Criteria:

* Systemic diseases associated with loss of periodontal supporting tissues.
* Metabolic bone diseases and systemic medications affecting bone metabolism.
* Craniofacial anomalies such as cleft lip and/or palate.
* Xerostomia.
* Tobacco-related habits such as smoking, tobacco chewing, etc.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Levels of ICTP in GCF and saliva samples before appliance placement, 24 hours, 3 days, 7 days, 14 days, and 21 days after archwire placement. | 21 days
  Measuring the Levels of collagen fragment ICTP in GCF and saliva samples before appliance placement, 24 hours, 3 days, 7 days, 14 days, and 21 days after archwire placement.
Levels of CTX in GCF and saliva samples before appliance placement, 24 hours, 3 days, 7 days, 14 days, and 21 days after archwire placement. | 21 days
  Measuring the Levels of collagen fragment CTX in GCF and saliva samples before appliance placement, 24 hours, 3 days, 7 days, 14 days, and 21 days after archwire placement.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Tareq, Principal Investigator — Principal Investigator
Locations (1):
- Alexandria university faculty of dentistry, Alexandria, Egypt